CLINICAL TRIAL: NCT03771196
Title: Clinical Evaluation of Bioactive Restorative vs. RMGI in Class V: A Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yehia Hafez Yehia, Yehia Hafez Yehia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7/12/2018
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Dental Restoration Failure
Keywords: Bioactive Restorative Material; ACTIVA Restorative; Resin Modified Glass Ionomer (RMGI); class V; Clinical perfomance
MeSH Terms: interventions — Fuji II LC cement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive-Restorative material (Experimental): Activa Bioactive-Restorative is an enhanced resin modified glass ionomer (RMGI) with an ionic resin matrix, a shock-absorbing resin component, and bioactive fillers that mimic the physical and chemical properties of natural teeth.
  Interventions: Other: Bioactive Restorative Material
- Resin Modified Glass Ionomer (RMGI) (Active Comparator): Fuji II Lc, fluoride-releasing restorative system that combines fluoride release of glass ionomer cement and acceptable esthetics a wear-resistant, self-adhesive, light-cured resin coating.
  Interventions: Other: Resin-modified glass ionomer

INTERVENTIONS:
Other: Bioactive Restorative Material — enhanced RMGIs with an ionic resin matrix, a shock-absorbing resin component, and bioactive fillers that mimic the physical and chemical properties of natural teeth
  Other Names: Activa Bioactive RestorActiva Bioactive Restorativeative
  Arms: Bioactive-Restorative material
Other: Resin-modified glass ionomer — Enhanced glass ionomer with acceptable mechanical properties and esthtic properties
  Other Names: Fuji II lc
  Arms: Resin Modified Glass Ionomer (RMGI)

SUMMARY:
Clinical performance of bioactive restorative material versus Resin Modifeid Glass Ionoer (RMGI) in class V o will be evaluated over 12 months using United State Public Health Criteria (USHPS) clinical criteria for the evaluation of direct and indirect restorations

DETAILED DESCRIPTION:
Recent developments in the province of material sciences, some novel materials require direct association with oral environment for renewal, recharging or enhancing of the constituents of the restoration to improve marginal integrity to decrease bacterial microleakage. Physical and chemical properties of dental restorations have been progressed such that individual components may exert a bioactive role in the prevention, remineralization, and restoration of active carious lesions.Fluoride containing restorative materials recently gained great attention. Fluoride decreases caries activity by being a bacteriostatic and by decreasing the solubility of enamel and dentin through its integration into tooth tissue to form fluoroapatite. Moreover, it aids to remineralize defected tooth structure after demineralization. conventional GICs and RMGICs are have high fluoride release and could be specified clinically to repair decayed non-biting areas in high caries risk patients.To enhance the mechanical properties of GIs, their constituents have been modified Comparatively, resin-modified GIs (RMGIs) with a longer working time, faster setting, higher early strength, and improved appearance and translucency. Unfortunately, the RMGI's mechanical properties of are different to resin composites. progressive development of material sciences has resulted in the introduction of bioactive restorative materials. These materials can activate a tissue repair mechanism for or synthesis and elicit a response from teeth and surrounding environment.

ELIGIBILITY:
Inclusion Criteria:

* Cervical Class V carious lesions.
* Age 18-50 years.
* Co-operative patients approving to participate in the study.
* Pulp asymptomatic vital carious posterior teeth.
* Presence of favorable occlusion and teeth are in normal contact with the adjacent teeth.

Exclusion Criteria:

* Systemic disease or severe medical complications.
* Allergic history concerning methacrylates
* Rampant caries
* Pregnancy
* Disabilities
* Heavy smoking; xerostomia
* Lack of compliance
* Evidence of severe bruxism, clenching, or temporomandibular joint disorders or bizarre habits

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in the clinical performance using United State Public Health Service (USHPS) | Change from the baseline at 6 months and12 months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] o ALKHUDHAIRY FI & ZH, A. 2016. Comparison of Shear Bond Strength and Microleakage of Various Bulk-fill Bioactive Dentin substitutes: An in vitro study. J Contemp Dent Pract, 17. o B. RANJBAR OMIDI, F. F. N., H. DEHGHAN, P. TAMIZ, M. MOHAMMADI SAVADROODBARI, AND R. JABBARIAN, 2018. Microleakage of an Enhanced Resin-Modified Glass Ionomer Restorative Material in Primary Molars. Journal of Dentistry of Tehran University of Medical Sciences (jdt), 15. o BANSAL, R., BURGESS, J. & LAWSON, N. C. 2016. Wear of an enhanced resin-modified glass-ionomer restorative material. Am J Dent, 29, 171-4. o CROLL, T. P., BERG, J. H. & DONLY, K. J. 2015. Dental repair material: a resin-modified glass-ionomer bioactive ionic resin-based composite. Compend Contin Educ Dent, 36, 60-5. o GAROUSHI, S., VALLITTU, P. K. & LASSILA, L. 2018. Characterization of fluoride releasing restorative dental materials. Dent Mater J, 37, 293-300. o HICKEL, R., PESCHKE, A., TYAS, M., MJOR, I., BAYNE, S., PETERS, M., HILLER, K. A., RANDALL, R., VANHERLE, G. & HEINTZE, S. D. 2010. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent, 12, 259-72. o MICHOU, S., LARSEN, L., BENETTI, A. R. & PEUTZFELDT, A. 2018. Adhesion and marginal integrity of bioactive restorative materials. Dental Materials, 34, e11. o NAGI, S. M., MOHARAM, L. M. & EL HOSHY, A. Z. 2018. Fluoride release and recharge of enhanced resin modified glass ionomer at different time intervals. Future Dental Journal. o NEMATOLLAHI, H., BAGHERIAN, A., GHAZVINI, K., ESMAILY, H. & MEHR, M. A. 2017. Microbial microleakage assessment of class V cavities restored with different materials and techniques: A laboratory study. Dental research journal, 14, 344-350. o OWENS, B. M., PHEBUS, J. G. & JOHNSON, W. W. 2018. Evaluation of the marginal integrity of a bioactive restorative material. Gen Dent, 66, 32-36. o PAMEIJER, C. H., GARCIA-GODOY, F., MORROW, B. R. & JEFFERIES, S. R. 2015. Flexural strength and flexural_fatigue. J Clin Dent, 26, 5. o PERDIGAO, J., DUTRA-CORREA, M., SARACENI, S. H., CIARAMICOLI, M. T. & KIYAN, V. H. 2012. Randomized clinical trial of two resin-modified glass ionomer materials: 1-year results. Oper Dent, 37, 591-601.2016. Guideline on Restorative Dentistry. Pediatr Dent, 38, 250-262.